CLINICAL TRIAL: NCT04546126
Title: Positron Emission Tomography (PET) Imaging of Cholesterol Trafficking: Clinical Evaluation of [18F]FNP-59 in Normal Human Subjects (Groups 2, 3 & 4)
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Benjamin Viglianti (Other)
Responsible Party: Sponsor-Investigator, Benjamin Viglianti, Assistant Professor of Radiology, University of Michigan
Organization: University of Michigan (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HUM00179097b
Record Dates: First submitted 2020-09-08; First posted 2020-09-11 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Radiotracer; Hypertension; Cholesterol
MeSH Terms: conditions — Hypertension | interventions — Dexamethasone; Cosyntropin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dexamethasone (Group 2) (Experimental): Participants will undergo an FNP-59 scan on day 0 in the am. Participants will then take
  1 mg dexamethasone 2x a day for 3 days to suppress cortisol production. Participants will then have a second FNP-59 scan on day 4 in the am.
  Interventions: Drug: Dexamethasone (Group 2); Combination Product: PET/CT Scan with FNP-59
- Cosyntropin (Group 3) (Experimental): Participants will undergo an FNP-59 scan on day 0 in the am. On day 4 the participant will arrive for imaging. Cosyntropin, 250 micro-gm will be administered IV. Five minutes following administration FNP-59 will be given. Following uptake of FNP-59 imaging will occur.
  Interventions: Drug: Cosyntropin (Group 3); Combination Product: PET/CT Scan with FNP-59
- Adrenal pathology (Group 4) (Experimental): Whole-body PET/CT scans will be done on 4 patients at 1 hr and the other 4 patients at 6 hours. All the patients will have a whole-body PET/CT scan at 3 hours.
  Interventions: Combination Product: PET/CT Scan with FNP-59

INTERVENTIONS:
Drug: Dexamethasone (Group 2) — Participants will take 1 mg dexamethasone 2x a day for 3 days to suppress cortisol production.
  Arms: Dexamethasone (Group 2)
Drug: Cosyntropin (Group 3) — Cosyntropin, 250 micro-gm will be administered IV. Five minutes following administration FNP-59 will be given. Following uptake of FNP-59 imaging will occur.
  Arms: Cosyntropin (Group 3)
Combination Product: PET/CT Scan with FNP-59 — FNP-59, a radiotracer, is administered for PET/CT scans.

SUMMARY:
This study will evaluate the feasibility of using a sub-therapeutic dose of a fluorine-18 analogue of NP-59 ([18F]FNP-59) to image the adrenal gland. Some participants are healthy normal subjects but have undergone interventions to manipulate hormones while other participants have known adrenal pathology.

DETAILED DESCRIPTION:
Groups 2 & 3 used hormone manipulation using information gathered from Group 1 which identified radiation dosimetry and optimal uptake time.

Group 4 (added to the study later) includes participants with known adrenal pathology. They will not have study associated hormone manipulation.

All groups will be given a radio-tracer and PET/CT scans.

The researchers believe that a fluorine-18 analogue of NP-59, [18F]FNP-59, would greatly improve the imaging characteristics, by providing a PET imaging cholesterol analogue with significantly improved radiation dosimetry, and improved localization / sensitivity / specificity without concern of thyroid exposure.

ELIGIBILITY:
Inclusion Criteria (Groups 2 & 3):

* Participants without any known adrenal pathology as normal controls for undergoing endocrine manipulation

Exclusion Criteria (Groups 2 & 3):

* Pregnancy
* Unable to do imaging
* Body weight greater than 400 lbs (181 Kg)
* Prisoners are not eligible
* Subjects unable to provide own consent are not eligible
* Current use of steroids, Oral contraceptives (OCP), spironolactone, estrogen, androgen, progesterone, Angiotensin-converting enzyme (ACE inhibitors)/ Angiotensin II receptor blockers (ARBs), or supplements that are hormone analogues.
* Known adrenal pathology

Inclusion Criteria (Group 4):

* Abnormal adrenal cortical hormone secretion

Exclusion Criteria (Group 4):

* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in [18F]FNP-59 chemistry uptake as measured by the standardized uptake value (SUV) based gland segmentation | Day 0, Day 4
  SUV will be reported. Both maximal and average SUVs will be calculated

SECONDARY OUTCOMES:
PET/CT image uptake score as measured by investigator visual assessment for each volume of interest (VOI) | Day 4
  Investigator scoring system (no increased uptake = 0, mild uptake = 1, moderate uptake = 2, high uptake = 3, relative to background. Higher scores indicate increased uptake.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin L Viglianti, M.D, Ph.D., Principal Investigator — University of Michigan
Locations (2):
- United States (2):
  - University of Michigan, Ann Arbor, Michigan
  - BAMF Health, Inc., Grand Rapids, Michigan

IPD SHARING:
Plan to Share IPD: No